CLINICAL TRIAL: NCT02623972
Title: A Phase 2 Study of Eribulin Followed by Doxorubicin and Cyclophosphamide as Preoperative Therapy for HER2-negative Inflammatory Breast Cancer
Brief Title: A Phase 2 Study of Eribulin Followed by AC as Preoperative Therapy for HER2-negative Inflammatory Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Filipa Lynce, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-292
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Breast Cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: inflammatory breast cancer; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — eribulin; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Eribulin > AC (Experimental): * Eribulin-Administered via iv, at predetermined dosage and schedule per cycle
  * Two research breast biopsies
  * Adriamycin (doxorubicin) via iv a predetermined dosage and schedule per cycle
  * Cyclophosphamide (AC) via iv a predetermined dosage and schedule per cycle
  * Surgical Removal of the breasts (Mastectomy) and axillary lymph node dissection
  * Radiation Therapy
  * Endocrine Therapy (if applicable)
  * Optional 5 Patient-Optional DCE-MRI (Dynamic Contrast Enhanced-Magnetic Resonance Imaging) scans
  Interventions: Drug: Eribulin; Drug: Adriamycin; Drug: Cyclophosphamide
- Arm B: AC > Eribulin (Experimental): * Adriamycin (doxorubicin) via iv a predetermined dosage and schedule per cycle
  * Cyclophosphamide (AC) via iv a predetermined dosage and schedule per cycle
  * Two research breast biopsies
  * Eribulin-Administered via iv, at predetermined dosage and schedule per cycle
  * Surgical Removal of the breasts (Mastectomy) and axillary lymph node dissection
  * Radiation Therapy
  * Endocrine Therapy (if applicable)
  * Optional 5 Patient-Optional DCE-MRI (Dynamic Contrast Enhanced-Magnetic Resonance Imaging) scans
  Interventions: Drug: Eribulin; Drug: Adriamycin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Eribulin — administered IV for 4 cycles
  Other Names: Halaven; B1939 mesylate
Drug: Adriamycin — administered IV with cyclophosphamide for 4 cycles
  Other Names: Doxorubicin
Drug: Cyclophosphamide — administered IV with adriamycin for 4 cycles
  Other Names: Cytoxan®; Neosar®

SUMMARY:
This research study is studying a drug called eribulin combined with standard treatment as a possible preoperative treatment for HER2 negative inflammatory breast cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

Eribulin works by interfering with cancer cell division, growth, and spread.

The goal of this research study is to evaluate inflammatory breast cancer's response to treatment with eribulin followed by AC chemotherapy (Cohort A) and also the response to treatment with AC followed by Eribulin (Cohort B) when given as a preoperative chemotherapy treatment for participants with HER2 negative inflammatory breast cancer.

ELIGIBILITY:
Inclusion Criteria:

-Participants must have histologically confirmed invasive breast cancer. All histologic subtypes are eligible.

-- Patients must NOT have HER2 positive status based on ASCO/CAP guidelines defined as: IHC 3+ based on circumferential membrane staining that is complete, intense and/or

FISH positive based on one of the three following criteria:

Single-probe average HER2 copy number ≥ 6.0 signals/cell; OR Dual-probe HER2/CEP17 ratio <2.0 with an average HER2 copy number ≥ 6.0 signals/cell; OR Dual-probe HER2/CEP17 ratio ≥2.0

* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of eribulin in participants <18 years of age, children are excluded from this study
* ECOG performance status ≤1 (Karnofsky ≥70%)
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal creatinine ≤1.5 × institutional upper limit of normal

    --- OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* Patients must have the clinical diagnosis of inflammatory breast cancer.
* Patients must be without evidence of visceral or bone involvement with metastatic cancer on physical exam or any diagnostic study. Extensive nodal involvement (distant or regional) is allowed.
* LVEF > 50% calculated by echocardiogram (ECHO)
* Patients may have bilateral breast cancer so long as one breast meets criteria for inflammatory breast cancer, and the breast with inflammatory breast cancer has never received prior therapy.
* The effects of eribulin on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of chemotherapy administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women of all races and ethnic groups are eligible for this trial. Because breast cancer predominantly affects females, it is anticipated that male enrollment will be < 5% of the overall study population.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to eribulin or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because eribulin is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with eribulin, breastfeeding should be discontinued if the mother is treated with eribulin. These potential risks may also apply to other agents used in this study.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with eribulin. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* A baseline corrected QT interval of > 470 ms.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Patients may not have received eribulin, paclitaxel, doxorubicin, or cyclophosphamide as anti-neoplastic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Lynce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Fanucci K, Yeh ED, Shi R, Qin L, Bay CP, DiLullo M, Patel A, Moore M, Herbert ZT, Harrison BT, Nakhlis F, Bellon J, Warren L, Guerriero JL, Tolaney SM, Regan M, Overmoyer B, Van Laere S, Lynce F. Neoadjuvant therapy with eribulin, doxorubicin and cyclophosphamide for patients with HER2-negative inflammatory breast cancer: a phase II study. Breast Cancer Res. 2025 Sep 29;27(1):171. doi: 10.1186/s13058-025-02108-4. PMID 41024110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2016 to December 2020
Groups:
- Arm A: Eribulin followed by AC: * Eribulin-Administered via iv, at predetermined dosage and schedule per cycle
  * Two research breast biopsies
  * Adriamycin (doxorubicin) via iv a predetermined dosage and schedule per cycle
  * Cyclophosphamide via iv a predetermined dosage and schedule per cycle
  * Surgical Removal of the breasts (Mastectomy) and axillary lymph node dissection
  * Radiation Therapy
  * Endocrine Therapy (if applicable)
  * Optional 5 Patient-Optional DCE-MRI (Dynamic Contrast Enhanced-Magnetic Resonance Imaging) scans
  Eribulin: administered IV for 4 cycles
  Adriamycin: administered IV with cyclophosphamide for 4 cycles
  Cyclophosphamide: administered IV with adriamycin for 4 cycles
- Arm B: AC followed by Eribulin: * Adriamycin (doxorubicin) via iv a predetermined dosage and schedule per cycle
  * Cyclophosphamide via iv a predetermined dosage and schedule per cycle
  * Two research breast biopsies
  * Eribulin-Administered via iv, at predetermined dosage and schedule per cycle
  * Surgical Removal of the breasts (Mastectomy) and axillary lymph node dissection
  * Radiation Therapy
  * Endocrine Therapy (if applicable)
  * Optional 5 Patient-Optional DCE-MRI (Dynamic Contrast Enhanced-Magnetic Resonance Imaging) scans
  Eribulin: administered IV for 4 cycles
  Adriamycin: administered IV with cyclophosphamide for 4 cycles
  Cyclophosphamide: administered IV with adriamycin for 4 cycles
Period: Overall Study
Arm/Group | Arm A: Eribulin followed by AC | Arm B: AC followed by Eribulin
Started | 16 | 6
Completed | 16 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Eribulin Followed by AC | Arm B: AC Followed by Eribulin | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Continuous [Median (Full Range); unit: years] — Age at enrollment
  years | 57 [35 to 64] | 59 [37 to 72] | 58 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 22
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 5 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 22
Estrogen Receptor Status [Count of Participants; unit: Participants] — <1% means negative, 1-10% means low positive, >10% means positive
  Participants
    <1% | 3 | 0 | 3
    1-10% | 0 | 1 | 1
    >10% | 13 | 5 | 18
Breast Cancer Stage [Count of Participants; unit: Participants] — Stage IIIB: The tumor has spread to the chest wall or caused swelling or ulceration of the breast, or it is diagnosed as inflammatory breast cancer.
  Stage IIIC: A tumor of any size that has spread to 10 or more axillary lymph nodes, the internal mammary lymph nodes, and/or the lymph nodes under the collarbone.
  Stage IV (metastatic): The tumor can be any size and has spread to other organs, such as the bones, lungs, brain, liver, distant lymph nodes, or chest wall
  Participants
    Unknown | 0 | 1 | 1
    IIIB | 14 | 3 | 17
    IIIC | 2 | 1 | 3
    IV | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Complete pathologic disease response (pCR) is defined as absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative therapy, based upon pathological assessment of surgical specimens. Those with invasive carcinoma present within the breast and axillary lymph nodes, and participants whose disease is not surgically resectable following preoperative treatment are considered as not having pCR.
Time Frame: Assessed after preoperative therapy with either 4 cycles of eribulin mesylate (3 wks) followed by 4 cycles of doxorubicin/cyclophosphamide (2 wks) or after 4 cycles of AC(2 wks) followed by 4 cycles of eribulin(3 wks). As such up to 20 weeks.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Eribulin followed by AC | Arm B: AC followed by Eribulin
Number analyzed (Participants) | 16 | 6
percentage of participants | 6.25 [0.66 to 22.22] | 0 [0 to 31.87]
Statistical Analysis 1: Comparison: Arm A: Eribulin followed by AC; Null Hypothesis: the proportion of participants experiencing pCR is ≤ 0.10, Alternative hypothesis that proportion pCR ≥ 0.30. Hypothesized False Positive Rate(α)=10%; Hypothesized False Negative Rate(1-β)=10%; Test type: Other; Simon minimax two-stage design; Pathelogic Complete Response Rate = 30 — Decision Rule: If the percentage of participants experiencing pathologic complete response (pCR) is ≤ 10% then the preoperative regimen is considered minimally effective. If the proportion of pCR ≥ 30% then the regimen is worthy of further study
Statistical Analysis 2: Comparison: Arm B: AC followed by Eribulin; Null Hypothesis: the proportion of participants experiencing pCR is ≤ 0.02, Alternative hypothesis that proportion pCR ≥ 0.23. Hypothesized False Positive Rate(α)=5%; Hypothesized False Negative Rate(1-β)=10%; Test type: Other; Simon minimax two-stage design; Pathelogic Complete Response Rate = 23 — Decision Rule: If the percentage of participants experiencing pathologic complete response (pCR) is ≤ 2% then the preoperative regimen is considered minimally effective. If the proportion of pCR ≥ 23% then the regimen is worthy of further study

2. Secondary Outcome: Disease Free Survival
Description: Disease-free survival (DFS) is defined for the participants who undergo surgery, as the duration of time from surgery until ipsilateral local-regional, contralateral or distant invasive recurrence or death from any cause; in the absence of an event, DFS will be censored at the date last know alive and free from recurrence.
Time Frame: DFS is assessed every cycle for 8 cycles. After protocol therapy, assessed every 3 months for 1 year, then every 6 months for 4 years, then annually until death.The DFS measurement duration is anticipated to last for at least 5 years.
Reporting Status: Not Posted, anticipated posting 2026-01

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) will be defined among all participants, as the duration of time from treatment initiation to a DFS event or progressive disease during preoperative therapy or treatment disease that is not surgically resectable; in the absence of an event, TTF will be censored at the date last know alive and free from recurrence or progression.
Time Frame: TTF is assessed every cycle for 8 cycles. After protocol therapy, assessed every 3 months for 1 year, then every 6 months for 4 years, then annually until death. The TTF measurement duration is anticipated to last for at least 5 years.
Reporting Status: Not Posted, anticipated posting 2026-01

4. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) will be defined two ways: among patients who undergo surgery, as time from surgery until death from any cause; and among all patients, as the time from treatment initiation until death from any cause. Censoring will use the date last known alive.
Time Frame: OS is assessed every cycle for 8 cycles. After protocol therapy, assessed every 3 months for 1 year, then every 6 months for 4 years, then annually until death. The OS measurement duration is anticipated to last for at least 5 years.
Reporting Status: Not Posted, anticipated posting 2026-01

5. Secondary Outcome: Residual Cancer Burden (RCB)
Description: Residual cancer burden is calculated and then categorized based on level of residual disease after neoadjuvant therapy and several other factors as assessed by pathologists.
  This method uses tumor size, the proportion of that tumor that is invasive carcinoma, the number of axillary lymph nodes containing metastatic carcinoma and the diameter of the largest metastasis in an axillary lymph node. This index is divided into 4 categories: RCB-0, RCB-I, RCB-II, and RCB-III.(RCB category "Unknown" if unable to determine RCB or missing data.) The previous categories are in order of increasing severity of RCB. Measurement of residual breast cancer burden can predict survival after neoadjuvant chemotherapy.
Time Frame: Assessed after preoperative therapy with either 4 cycles of eribulin mesylate (3 wks) followed by 4 cycles of doxorubicin/cyclophosphamide (2 wks) or after 4 cycles of AC(2 wks) followed by 4 cycles of eribulin(3 wks). As such summed up to 20 weeks.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Eribulin followed by AC | Arm B: AC followed by Eribulin
Number analyzed (Participants) | 16 | 6
percentage of participants
  RCB-0 | 6.25 [0.66 to 22.22] | 0 [0 to 31.87]
  RCB-I | 12.5 [3.37 to 29.96] | 0 [0 to 31.87]
  RCB-II | 25 [11.38 to 43.89] | 50 [20.09 to 79.91]
  RCB-III | 56.25 [37.5 to 73.71] | 33.33 [9.26 to 66.68]
  Unknown | 0 [0 to 13.4] | 16.67 [1.74 to 51.03]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality measurement is anticipated to last for at least 5 years. It is assessed every cycle for 8 cycles during treatment. After protocol therapy, every 3 months for 1 year, then every 6 months for 4 years, then annually until death. Adverse events(SAEs and OAEs) are assessed every cycle for 8 cycles. After protocol therapy, assessed approximately 4 weeks following completion of therapy. The median(range) number of competed cycles of therapy was 8(7-8). As such up to 24 weeks.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Arm A: Eribulin followed by AC | Arm B: AC followed by Eribulin
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/16 | 1/6
Other Adverse Events (participants affected / at risk) | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin followed by AC (N=16) | Arm B: AC followed by Eribulin (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Eribulin followed by AC (N=16) | Arm B: AC followed by Eribulin (N=6)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 10 | 5
Vomiting (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders and administration site conditions) | 1 | 0
Fatigue (General disorders and administration site conditions) | 15 | 6
Flu like symptoms (General disorders and administration site conditions) | 1 | 0
Pain (General disorders and administration site conditions) | 2 | 2
Fever (General disorders and administration site conditions) | 0 | 2
Papulopustular rash (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 3 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 4
Neutrophil count decreased (Investigations) | 3 | 0
Weight loss (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 7 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 3
Tremor (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flashes (Vascular disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02623972/Prot_SAP_000.pdf